CLINICAL TRIAL: NCT01034423
Title: Omega-3 Fatty Acids and Health Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Stine Marie Ulven, Associate Professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 6.2008.2215
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Focus: health effects from omega-3 fatty acids, from fish oil with different quality
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- omega-3 high quality (Experimental)
  Interventions: Dietary Supplement: Omega-3; Dietary Supplement: sun flower oil
- omega-3 low quality (Experimental)
  Interventions: Dietary Supplement: Omega-3; Dietary Supplement: sun flower oil
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Omega-3; Dietary Supplement: sun flower oil

INTERVENTIONS:
Dietary Supplement: Omega-3 — Capsules with omega-3 fatty acids.
Dietary Supplement: sun flower oil — Capsules with sun flower oil.

SUMMARY:
The investigators want to study health effects from omega-3 fatty acids, from fishoil with different quality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals.

Exclusion Criteria:

* Pregnant women, lactating women, chronic diseases and smoking.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Primary and secondary oxidation products | baseline (0 weeks), 3 weeks and 7 weeks

SECONDARY OUTCOMES:
inflammatory markers | after 0,3 and 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stine M Ulven, PhD, Study Chair — Oslo Metropolitan University

REFERENCES:
- [Derived] Myhrstad MC, Ottestad I, Gunther CC, Ryeng E, Holden M, Nilsson A, Bronner KW, Kohler A, Borge GI, Holven KB, Ulven SM. The PBMC transcriptome profile after intake of oxidized versus high-quality fish oil: an explorative study in healthy subjects. Genes Nutr. 2016 May 31;11:16. doi: 10.1186/s12263-016-0530-6. eCollection 2016. PMID 27551317
- [Derived] Myhrstad MC, Ulven SM, Gunther CC, Ottestad I, Holden M, Ryeng E, Borge GI, Kohler A, Bronner KW, Thoresen M, Holven KB. Fish oil supplementation induces expression of genes related to cell cycle, endoplasmic reticulum stress and apoptosis in peripheral blood mononuclear cells: a transcriptomic approach. J Intern Med. 2014 Nov;276(5):498-511. doi: 10.1111/joim.12217. Epub 2014 Mar 20. PMID 24641624
- [Derived] Ottestad I, Hassani S, Borge GI, Kohler A, Vogt G, Hyotylainen T, Oresic M, Bronner KW, Holven KB, Ulven SM, Myhrstad MC. Fish oil supplementation alters the plasma lipidomic profile and increases long-chain PUFAs of phospholipids and triglycerides in healthy subjects. PLoS One. 2012;7(8):e42550. doi: 10.1371/journal.pone.0042550. Epub 2012 Aug 28. PMID 22952598
- [Derived] Ottestad I, Vogt G, Retterstol K, Myhrstad MC, Haugen JE, Nilsson A, Ravn-Haren G, Nordvi B, Bronner KW, Andersen LF, Holven KB, Ulven SM. Oxidised fish oil does not influence established markers of oxidative stress in healthy human subjects: a randomised controlled trial. Br J Nutr. 2012 Jul;108(2):315-26. doi: 10.1017/S0007114511005484. Epub 2011 Dec 5. PMID 22136711